# <u>Can You Reduce Diabetes Symptomatology by Becoming Your 'Best Possible Self'?: The Role of Stress and Resilience</u>

Study Protocol and Statistical Analysis Plan

Last Edited: 14/09/2018

#### Protocol

<u>Title: Can You Reduce Diabetes Symptomatology by Becoming Your 'Best Possible Self'?: The Role of Stress and Resilience.</u>

## **Research Question**

How does the 'Best Possible Self' Task influence stress and resilience when used as a diabetes prevention tool?

## **Background**

Diabetes mellitus continues to be a global burden and it affects millions of people around the world (Bommer et al., 2017). Prevalence figures from 2015 revealed that approximately 5 million adults in England alone were at high risk of developing type 2 diabetes specifically (Public Health England, 2016), a form of the disease that is largely preventable via lifestyle changes (Klein, Sheard, Pi-Sunyer, Daly, Wylie-Rosett, Kulkarni, & Clark, 2004). Typically, education interventions are utilised in efforts to promote awareness and generate behavioural change prior to formal diagnosis (Lian, McGhee, Chau, Wong, Lam, & Wong, 2017; Roberts, Barry, Craig, Airoldi, Bevan, & Greenhalgh, 2017) but this is not always enough to motivate individuals to act (Horigan, Davies, Findlay-White, Chaney, & Voates, 2017). Research has demonstrated that emotionality plays a significant role not only in lifestyle change but also in symptom management (Rasmussen, Smith, Maxson, Bernard, Cha, Agerter, & Shah, 2013). Experiencing mental illness, distress, or even just a high frequency of negative emotions can negatively influence dieting and exercising behaviours (Ciechanowski, Katon, & Russo, 2000), for example, increasing risk. However, novel findings have shown that experiencing positive emotions (such as happiness, optimism, interest, feelings of strength, etc.) can have the opposite effect and may help empower the individual to make the changes they need to improve their health (Garland, Fredrickson, Kring, Johnson, Meyer, & Penn, 2010). Interventions designed to foster positive emotions specifically are in development across psychology and have shown to improve mental as well as physical health outcomes (Chew, Vos, Heijmanns, Metzendorf, Scholten, & Rutten, 2015). This has been supported by our own investigations whereby we discovered that one such "positive" intervention reduces certain diabetes symptoms regardless of the individual's level of risk.

The positive intervention we have been using is an adapted version of the 'Best Possible Self' (BPS) task – a goal setting exercise that has shown to be effective in improving illness management and facilitating positive emotions (King, 2001). Its influence on diabetes symptoms is a novel finding, and with this study we are hoping to further investigate how it achieves this effect. According to the Stress Buffering Model of Physical Activity (Pressman & Cohen, 2005), psychological stress is the catalyst that triggers behavioural and physiological responses critical to health and positive emotions improve health by helping people to cope. The Broaden and Build Theory of Positive Emotions, meanwhile, suggests that this is because positive emotions allow people to build resilience (Fredrickson, 2001). Research around stress and resilience has shown these factors to be important not only in physical health of people with diabetes (Yi, Vitaliano, Smith, Yi, & Weinger, 2008) but for also decreasing illness symptomatology in non-clinical samples more generally (Steinhardt & Dolbier, 2008). As such, this proposed study aims to assess the role that stress and resilience may play in mediating the relationship between BPS and diabetes symptomatology.

#### <u>Hypotheses:</u>

The 'Best Possible Self' task will increase resilience and alleviate stress in order to reduce symptoms of diabetes in a non-clinical sample.

# Methodology

See flowchart below:

# **Study Created**

Following ethical approval, study is created and set up on Qualtrics, an online survey system.

# **Study Advertised**

Bulk Emails, Social Media, SONA, Public Forums.

## **Participants Recruited**

Interested individuals will be provided with an information sheet, the opportunity to ask questions, and a link to the study where they can provide consent.

# **Participants Randomised**

150+ participants are then randomised into one of two conditions on Qualtrics.

#### **Intervention Group**

Participants receive the BPS straight away.

#### Control

Participants are told they are on a waiting list to receive the BPS at the end of the study period.

# **Time Point 1 Questionnaires**

All participants then complete CANRISK (diabetes risk), PSS (stress), 6BRS (resilience), and DSC-R (diabetes symptoms) questionnaires.

# 4-week interval

# **Time Point 2 Questionnaires**

Participants return to Qualtrics and repeat PSS, 6BRS, and DSC-R.

## <u>Debrief</u>

#### <u>Analysis</u>

A series of MANOVAs will be used to assess the influence of the BPS on diabetes symptoms over time and across groups. MANCOVAs will be used to control for diabetes risk. A mediation analysis will be conducted using the PROCESS software (Hayes, 2012) to assess whether the relationship between the BPS and diabetes symptoms is mediated by stress and resilience.



## References

Bommer, C. Heesemann, E., Sagalova, V., Manne-Goehler, J., Atun, R., Barnighausen, T., & Vollmer, S. (2017). The global economic burden of diabetes in adults aged 20-79 years: A cost-of-illness study. *The Lancet Diabetes & Endocrinology*, *5*(6), 423-430.

Chew, B. H., Vos, R., Heijmans, M., Metzendorf, M. I., Scholten, R. J., & Rutten, G. E. (2015). Psychological interventions for diabetes-related distress in adults with type 2 diabetes mellitus. *The Cochrane Library*.

Ciechanowski, P. S., Katon, W. J., & Russo, J. E. (2000). Depression and diabetes: Impact of depressive symptoms on adherence, function, and costs. *Archives of Internal Medicine*, *160*(21), 3278-3285.

Fredrickson, B. L. (2001). The role of positive emotions in positive psychology: The broaden-and-build theory of positive emotions. *American Psychologist*, *56*(3), 218.

Garland, E. L., Fredrickson, B., Kring, A. M., Johnson, D. P., Meyer, P. S., & Penn, D. L. (2010). Upward spirals of positive emotions counter downward spirals of negativity: Insights from the broaden-and-build theory and affective neuroscience on the treatment of emotion dysfunctions and deficits in psychopathology. *Clinical Psychology Review*, *30*(7), 849-864.

Hayes, A. F. (2012). PROCESS: A versatile computational tool for observed variable mediation, moderation, and conditional process modelling.

Horigan, G., Davies, M., Findlay-White, F., Chaney, D., & Coates, V. (2017). Reasons why patients referred to diabetes education programmes choose note to attend: A systematic review. *Diabetes Medicine*, *34*(1), 14-26.

King, L. A. (2001). The health benefits of writing about life goals. *Personality and Social Psychology Bulletin,* 27(7), 798-807.

Klein, S., Sheard, N., F., Pi-Sunyer, X., Daly, A., Wylie-Rosett, J., Kulkarni, K., & Clark, N. G. (2004). Weight management through lifestyle modification for the prevention and management of type 2 diabetes: Rationale and strategies. *Diabetes Care, 27*(8), 2067-2073.

Lian, J. X., McGhee, S. M., Chau, J., Wong, C. K. H., Lam, C. L. K., & Wong, W. C. W. (2017). Systematic review on the cost-effectiveness of self-management education programme for type 2 diabetes mellitus. *Diabetes Research and Clinical Practice*, 127, 21-34.

Pressman, S. D., & Cohen, S. (2005). Does positive affect influence health? *Psychological Bulletin, 131*(6), 925.

Public Health England (2015). Analysis of non-diabetes hyperglycaemia prevalence in England (Press Release). Retrieved from <a href="https://www.gov.uk/government/publications/nhs-diabetes-prevention-programme-non-diabetic-hyperglycaemia">https://www.gov.uk/government/publications/nhs-diabetes-prevention-programme-non-diabetic-hyperglycaemia</a>.

Rasmussen, N. H., Smith, S. A., Maxson, J. A., Bernard, M. E., Cha, S. S., Agerter, D. C., & Shah, N. D. (2013). Association of HbA1c with emotion regulation, intolerance of uncertainty, and purpose in life in type 2 diabetes mellitus. *Primary Care Diabetes*, 7(3), 213-221.

Roberts, S., Barry, E., Craig, D., Airoldi, M., Bevan, G., & Greenhalgh, T. (2017). Preventing type 2 diabetes: Systematic review of studies of cost-effectiveness of lifestyle programmes and metformin, with and without screening, for pre-diabetes. *BMJ Open, 7*(11), e017184.

Steinhardt, M., & Dolbier, C. (2008). Evaluation of a resilience intervention to enhance coping strategies and protective factors and decrease symptomatology. *Journal of American College Health*, *56*(4), 445-453.

Yi, J. P., Vitaliano, P. P., Smith, R. E., Yi, J. C., & Weinger, K. (2008). The role of resilience on psychological adjustment and physical health in patients with diabetes. *British Journal of Health Psychology*, 13(2), 311-325.